CLINICAL TRIAL: NCT00088543
Title: Pilot Trial of Two Dose Levels of Thymoglobulin as Part of a Myeloablative-Conditioning for a Human Leukocyte Antigen (HLA) Identical Matched Related Donor (MRD) Stem Cell Transplant (SCT) With Cyclosporine (CSa) as Post-transplant Graft vs. Host Disease (GvHD) Prophylaxis
Brief Title: Thymoglobulin to Prevent Acute Graft vs. Host Disease (GvHD) in Patients With Acute Lymphocytic Leukemia (ALL) or Acute Myelogenous Leukemia (AML) Receiving a Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SMC-101-1026
Record Dates: First submitted 2004-07-29; First posted 2004-07-30 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myelogenous Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Graft vs. Host Disease (GvHD)
Keywords: Acute myelogenous leukemia (AML); Acute lymphocytic leukemia (ALL); Anti-T cell antibodies; Allogenic stem cell transplant; Graft vs. Host Disease (GvHD)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Graft vs Host Disease | interventions — thymoglobulin; Antilymphocyte Serum

ARMS (2):
- 1 Low dose (Experimental): total dose 4.5 mg/kg Thymoglobulin
  Interventions: Biological: Thymoglobulin [Anti-Thymocyte Globulin (Rabbit)]
- 2 High dose (Experimental): total dose 8.5 mg/kg Thymoglobulin
  Interventions: Biological: Thymoglobulin [Anti-Thymocyte Globulin (Rabbit)]

INTERVENTIONS:
Biological: Thymoglobulin [Anti-Thymocyte Globulin (Rabbit)] — total dose 4.5 mg/kg
  Arms: 1 Low dose
Biological: Thymoglobulin [Anti-Thymocyte Globulin (Rabbit)] — total dose 8.5 mg/kg
  Arms: 2 High dose

SUMMARY:
This study involves the use of a drug called Thymoglobulin, which is approved in the USA to treat kidney transplant rejection and in Canada to treat and to prevent kidney transplant rejection. Thymoglobulin is not approved for the treatment or prophylaxis of graft versus host disease in bone marrow transplantation. This study is to evaluate two (2) doses of Thymoglobulin and its safety and effectiveness when used with a "myeloablative" conditioning regimen prior to receiving a stem cell transplant (also called bone marrow transplantation) from a matched, related donor.

A myeloablative regimen is typically composed of chemotherapy and radiation and destroys the subject's existing bone marrow.

Subjects meeting all inclusion and exclusion criteria and who have a relative with matching (genetically similar) stem cells who are also willing to donate them (i.e. matched-related-donor) are eligible to participate in this study. Following myeloablative therapy, the donor's cells are then transplanted (i.e. infused) into the subject's blood stream.

One of the most common complications of this type of transplant is graft-versus-host disease (GvHD). This is a condition where the transplanted donor cells attack the transplant recipient's body. Treatments, such as cyclosporine, are used to minimize the risk of GvHD following stem cell transplantation.

To enter this study, subjects must be having a matched-related donor stem cell transplant. If a subject qualifies for entry into this study, he/she will be assigned to receive Thymoglobulin at a dose of 4.5 mg/kg or 8.5 mg/kg. The treatment assignment is random and is not chosen by the subject or their physician.

Subjects are admitted to the hospital for the transplant procedure and are treated with Thymoglobulin over 3-5 days just prior to receiving the donor stem cells. The subject will also receive standard GvHD prophylaxis with cyclosporine. Methotrexate, which is commonly used by transplant centers to minimize the risk of GvHD, will not be used in this study.

Subjects will be monitored during treatment with Thymoglobulin and during the transplant hospitalization. Additional subject monitoring occurs at month 1, 100 days and 6 months following the transplant.

Approximately 60 study subjects from approximately 14 transplant centers in the United States and Canada will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an HLA-A, -B and -DRB1 identical related donor and must be fully matched at Class II. A high resolution molecular HLA typing (at least 4 digits) is mandatory for HLA Class II and optional for HLA Class I
* Subject has confirmed diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) with acute myeloid leukemia (including secondary leukemia) in first complete remission (CR2) or acute lymphoid in CR1 or CR2.
* Subject is >= 18 and <= 55 years of age.
* Subject is receiving a myeloablative-conditioning regimen
* Men and women of childbearing age potential agree to practice an acceptable and reliable form of contraception during the study. Women must not be lactating or pregnant, and must have a negative serum pregnancy test.
* Subject has been fully informed and has signed an IRB-approved informed consent form.
* Subject is willing and able to follow study procedures for the 6 months post-transplant.
* The subject must be serologically negative for human immunodeficiency virus (HIV).
* Subject agrees to be followed for possible long-term safety outcomes for up to 12 months post-transplant.
* Subject has an ECOG performance score of 0-2.
* Subject has a creatinine of < 2.0mg/dL or creatinine clearance of > 50mL/min.
* Subject has an ejection fraction of >= 40%
* Subject has a serum bilirubin of < 2mg/dL.

Exclusion Criteria:

* Subject is receiving fludarabine, a non-myeloablative regimen, or other purine analogues as part of the conditioning regimen.
* Subject is receiving an ex vivo engineered or processed graft (CD34+ enrichment, T-cell depletion, etc.)
* Subject has documented uncontrolled central nervous system (CNS) disease.
* Subject is expected to receive or has received methotrexate for GvHD prophylaxis.
* Subject has alanine aminotransferase (ALT)or aspartate aminotransferase (AST) level of > 3x the upper limit of normal range within 3 weeks prior to transplant.
* Subject has used any experimental agent within 30 days prior to the date of signing the informed consent.
* Subject is receiving or has received a bone marrow transplant from a donor who has positive serology for HIV, hepatitis B virus(HBV), hepatitis C virus (HCV) or syphilis.
* Subject has a known contraindication to administration of rabbit anti-thymocyte globulin.
* Subject is currently abusing drugs or alcohol or, in the opinion of the Investigator, is at high risk for poor compliance.
* Subject, who in the opinion of the Investigator, has significant medical or psychological problems that warrants exclusion. Examples of significant problems include, but are not limited to, morbid obesity or severe cardiac disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade II to IV acute GvHD in the first 100 days after transplant. | 100 days

SECONDARY OUTCOMES:
Incidence of treatment related adverse events and serious adverse events at 100 days and 6 months post transplant | 100 days and 6 months
Patient survival at 100 days and 6 months after transplant | 100 days and 6 months
transplant related mortality at 100 days or 6 months after transplant | 100 days and 6 months
severity and outcomes of acute GvHD | 100 days & 6 mos
any events of infection at 100 days and 6 months after transplant | 100 days and 6 months
incidence (or absence) of mucositis | continuous
how many days in the first month after transplant certain types of narcotics are used to reduce pain | 30days
whether the subject's blood counts after transplant reach a stable level and how quickly | Continuous
incidence of re-hospitalization in the first 6 months after transplant | 6 months
any recurrence of the subject's leukemic disease, and how long the subject was able to stay in remission | Continuous
incidence and severity of chronic GvHD, and the extent, after 100 days and 6 months after transplant | 100 days and 6 months
Disease free survival | 100 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (14):
- United States (12):
  - University of Alabama-Birmingham Hospital, Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - Shands at the University of Florida, Division of Hematology/Oncology, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital Cox Bldg Room 640, Boston, Massachusetts
  - Dana Farber Cancer Institute Dana 1B11, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center KS121, Brookline, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, University Health Network, Toronto, Ontario

REFERENCES:
- See also: US FDA Approved Full Prescribing Information for Thymoglobulin® — http://www.thymoglobulin.com/home/thymo_pdf_pi.pdf